CLINICAL TRIAL: NCT05829980
Title: Contoura Topography-guided Ablation Versus Wavefront-optimized Ablation for Correction of Astigmatism
Brief Title: Contoura vs Wavefront Optimized Ablation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hebatallah MT Abdelmoniem (Other)
Responsible Party: Sponsor-Investigator, Hebatallah MT Abdelmoniem, Assistant Lecturer, Assiut University
Organization: Assiut University (Other)
Other Study IDs: CONvsWFO
Record Dates: First submitted 2023-04-13; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Astigmatism
Keywords: Contoura; Wavefront optimized ablation; LASIK; PRK
MeSH Terms: conditions — Astigmatism | interventions — Keratomileusis, Laser In Situ; Photorefractive Keratectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group A: Contoura topography-guided LASIK
  Interventions: Procedure: Laser assisted in-situ keratomileusis
- Group B: Contoura topography-guided PRK
  Interventions: Procedure: Photorefractive keratectomy
- Group C: Wavefront-optimized LASIK
  Interventions: Procedure: Laser assisted in-situ keratomileusis
- Group D: Wavefront-optimized PRK
  Interventions: Procedure: Photorefractive keratectomy

INTERVENTIONS:
Procedure: Laser assisted in-situ keratomileusis — Laser-Assisted In Situ Keratomileusis is a procedure that permanently changes the shape of the cornea using an excimer laser and the mechanical microkeratome (a blade device) used to cut a flap in the cornea.
  Other Names: LASIK
  Groups: Group A; Group C
Procedure: Photorefractive keratectomy — Photorefractive keratectomy is a laser refractive procedure used to ablate the corneal stroma to correct refractive errors without cutting flap
  Other Names: PRK
  Groups: Group B; Group D

SUMMARY:
To evaluate the efficacy, safety and accuracy of Contoura topography-guided LASIK & PRK in comparison to Wavefront optimized LASIK & PRK in virgin eyes with astigmatism.

DETAILED DESCRIPTION:
In Upper Egypt, The second principal cause of blindness was uncorrected refractive errors accounting for 16% of sample population. It was reported that astigmatism (defined as cylinder power > 0.5 D) was the most common refractive errors in children and adults followed by hyperopia and myopia.

Laser vision correction has been established over the last 2 decades as a safe and effective intervention to treat refractive errors, being one of the main techniques practiced globally.

However, many subjects after LASIK had uncorrected distance visual acuity (UDVA) greater than 1.0, they complain about poor night vision, glare, and double vision. As studies have shown that every 1° deviation of the astigmatic axis could result in loss of correction of 3.3%. Even residual astigmatism less than 0.50D could have an actual impact on visual quality.

Excimer laser ablation used in the correction of refracted errors especially astigmatism may reduce quality of vision, and that is attributed to the induced optical aberrations. The most prevalent of these optical aberrations is the spherical aberration.

Among multiple sophisticated profiles that developed to optimize visual outcomes, wavefront optimized profile which compensate for corneal curvature to reduce spherical aberration.

The topographic guided profiles which consider the shape of the anterior corneal surface. Contoura topography guided ablation corrects astigmatic power and axis to create a more uniform, aberration-free cornea.

Treating astigmatism can be challenging as the conventional patterns of Excimer laser treatment of astigmatism is known to be less predictable than that of spherical refractive errors.

ELIGIBILITY:
Inclusion Criteria:

* Astigmatism (up to 5.0 diopters) or less.
* Central corneal thickness (CCT) of 500 microns or more
* Estimated Residual stromal bed thickness (RSB) of 280 microns or more
* Subject has provided written informed consent

Exclusion Criteria:

* Keratoconus
* Abnormal topography
* previous ocular trauma or eye surgery
* pre-existing diseases of the vitreous, macula, or optic nerve that can affect visual outcome
* patients with uveitis and anterior segment pathology
* patients with corneal pathology or Severe dry eye
* pregnancy or breast-feeding females
* uncontrolled vascular or autoimmune disease

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: participants who are candidates and scheduled for excimer laser treatment either LASIK or PRK
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Change in Postoperative UDVA compared to preoperative CDVA (in LogMAR) | 3 month
  UCVA 3 month after surgery compared to baseline preoperative CDVA
Number of lines of preoperative CDVA compared to postoperative | 3 month
  Change in lines of CDVA from baseline preoperative to 3 month postoperative (in LogMAR)
Amount of Residual Astigmatism postoperatively (in Diopters) | 3 month
  residual astigmatism 3 month postoperatively
Postoperative mean spherical equivalent MSE compared to Preoperative MSE (in Diopters) | 3 month
  changes in mean spherical equivalent baseline preoperative to 3 month postoperative

SECONDARY OUTCOMES:
Change in Contrast sensitivity test | 3 month
Amount of High order aberrations | 3 month
  (Spherical aberration, trefoil, vertical & horizontal coma)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A. Sayed, Ass. Prof., Study Chair — Assiut University

REFERENCES:
- [Background] Mousa A, Courtright P, Kazanjian A, Bassett K. Prevalence of visual impairment and blindness in Upper Egypt: a gender-based perspective. Ophthalmic Epidemiol. 2014 Jun;21(3):190-6. doi: 10.3109/09286586.2014.906629. Epub 2014 Apr 18. PMID 24746251
- [Background] Hashemi H, Fotouhi A, Yekta A, Pakzad R, Ostadimoghaddam H, Khabazkhoob M. Global and regional estimates of prevalence of refractive errors: Systematic review and meta-analysis. J Curr Ophthalmol. 2017 Sep 27;30(1):3-22. doi: 10.1016/j.joco.2017.08.009. eCollection 2018 Mar. PMID 29564404
- [Background] Lukenda A, Martinovic ZK, Kalauz M. Excimer laser correction of hyperopia, hyperopic and mixed astigmatism: past, present, and future. Acta Clin Croat. 2012 Jun;51(2):299-304. PMID 23115960
- [Background] Bailey MD, Zadnik K. Outcomes of LASIK for myopia with FDA-approved lasers. Cornea. 2007 Apr;26(3):246-54. doi: 10.1097/ICO.0b013e318033dbf0. PMID 17413947
- [Background] Lin Y, Su HJ, Yuan MZ, Zhang Y. Vector analysis of Contoura Vision for the correction of myopia and myopic astigmatism. Int J Ophthalmol. 2022 Jun 18;15(6):983-989. doi: 10.18240/ijo.2022.06.17. eCollection 2022. PMID 35814884
- [Background] Villegas EA, Alcon E, Artal P. Minimum amount of astigmatism that should be corrected. J Cataract Refract Surg. 2014 Jan;40(1):13-9. doi: 10.1016/j.jcrs.2013.09.010. PMID 24355718
- [Background] Gatinel D, Malet J, Hoang-Xuan T, Azar DT. Analysis of customized corneal ablations: theoretical limitations of increasing negative asphericity. Invest Ophthalmol Vis Sci. 2002 Apr;43(4):941-8. PMID 11923232
- [Background] Kanellopoulos AJ. Topography-modified refraction (TMR): adjustment of treated cylinder amount and axis to the topography versus standard clinical refraction in myopic topography-guided LASIK. Clin Ophthalmol. 2016 Nov 3;10:2213-2221. doi: 10.2147/OPTH.S122345. eCollection 2016. PMID 27843292
- [Background] Motwani M. The use of WaveLight(R) Contoura to create a uniform cornea: the LYRA Protocol. Part 3: the results of 50 treated eyes. Clin Ophthalmol. 2017 May 16;11:915-921. doi: 10.2147/OPTH.S133841. eCollection 2017. PMID 28553071
- [Background] Canones-Zafra R, Katsanos A, Garcia-Gonzalez M, Gros-Otero J, Teus MA. Femtosecond LASIK for the correction of low and high myopic astigmatism. Int Ophthalmol. 2022 Jan;42(1):73-80. doi: 10.1007/s10792-021-02001-x. Epub 2021 Aug 9. PMID 34370173